CLINICAL TRIAL: NCT02816359
Title: Impact of Patient Position on the Value of Esophageal Pressure. pEsition Study.
Brief Title: Position and Esophageal Pressure
Acronym: pEsition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL16_0152
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Position patient; Esophageal pressure
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- head-bed position (Other): Head-bed position at 0° for 30 minutes then head-bed position at 30° for 30 minutes
  Interventions: Other: head-bed position

INTERVENTIONS:
Other: head-bed position — Head-bed position at 0° for 30 minutes then head-bed position at 30° for 30 minutes

SUMMARY:
Esophageal pressure measurements are used in moderate/severe Accurate Respiratory Distress SyndromeARDS patients in order to set ventilator settings. There might be variations of the measured value according to the patient position (0° vs 30°) at the time of measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Acute respiratory failure defined by PaO2/FIO2< 300 mmHg or pH<7,35 and pCO2>45mmHg or Moderate or severe Accurate Respiratory Distress Syndrome ARDS defined by:

  * New or worsening respiratory symptoms in the previous week.
  * Bilateral opacities-not fully explained by effusions, lobar/lung collapse, or Nodules
  * Respiratory failure not fully explained by cardiac failure or fluid overload
  * PaO2/FIO2< 200 mmHg and PEEP ≥ 5 cm H2O and VT ≤6 ml/kg of Ideal Body Weight
* Patient intubated or tracheotomized and receiving mechanical ventilation
* Indication of esophageal measurement decided by the clinician

Exclusion Criteria:

* Contraindication to naso-gastric tube insertion :

  * Recent gastro-duodenal ulcer
  * Stage III esophageal varices
* Refractory intracranial hypertension
* Unstabilized spine fracture
* Surgical contraindication
* Burns on more than 20 % of the body surface
* Underlying disease with a life expectancy of less than one year
* End-of-life decision before inclusion
* Pregnant or breast-feeding patients
* Subject deprived of freedom, minor, subject under a legal protective measure
* Research team unavailability
* Lack of medical care plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Total End-expiratory esophageal pressure | 30min after change of position
  After end-expiratory pause on the ventilator, absolute value of the esophageal pressure is measured (in Head-bed position at 30° then in head-bed position at 0° )

SECONDARY OUTCOMES:
End-inspiratory esophageal pressure | 30min after change of position
  After end-inspiratory pause on the ventilator, absolute value of the esophageal pressure is measured (in Head-bed position at 30° then in head-bed position at 0° )
Gastric pressure | 30min after change of position
  After end-expiratory pause and end-inspiratory pause on the ventilator, absolute value of the gastric pressure is measured (in Head-bed position at 30° then in head-bed position at 0° )
End-expiratory lung volume | 30min after change of position
  End-expiratory lung volume is measured with nitrogen wash-in wash-out method, available in the ventilator (in Head-bed position at 30° then in head-bed position at 0° )

CONTACTS AND LOCATIONS:
Overall Officials: Claude Guerin, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Croix-Rousse, Lyon, France

REFERENCES:
- [Result] Mezidi M, Guerin C. Effect of body position and inclination in supine and prone position on respiratory mechanics in acute respiratory distress syndrome. Intensive Care Med. 2019 Feb;45(2):292-294. doi: 10.1007/s00134-018-5493-1. Epub 2018 Dec 7. No abstract available. PMID 30535985